CLINICAL TRIAL: NCT04090814
Title: Transcutaneous Electrical Nerve Stimulation Reduces Movement-Evoked Pain in People With Chronic Low Back Pain: A Randomised Crossover Study
Brief Title: TENS Reduces Movement-Evoked Pain in People With CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Lynn Leemans, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LLeemans
Record Dates: First submitted 2019-09-05; First posted 2019-09-16 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Movement-Evoked Pain during TENS treatment (Experimental): Participants performed several physical tasks while using the HeatTens device (HV-F311-E). During these tasks, participants needed to rate their pain.
  Interventions: Device: HeatTens (HV-F311-E)
- Movement-Evoked Pain (No Intervention): Participants performed several physical tasks during with their pain was assessed.

INTERVENTIONS:
Device: HeatTens (HV-F311-E) — (1) 2~108 Hertz (modulation program inside); (2) 100 microseconds (pulse duration)
  Arms: Movement-Evoked Pain during TENS treatment

SUMMARY:
In this cross-over study 25 patients with chronic low back pain (CLBP) were tested for pain relief in 2 conditions: while using the Transcutaneous Electrical Nerve Stimulation (TENS) application and without using it. Primary outcome: Movement-Evoked Pain (MEP). This was measured using the Back Performance Scale (BPS) and a 5-minute walk test (5MWT). Participants performed 5 functional tasks and were asked to rate their pain before, during, and after each movement on a numeric rating score scale. The same principle will be used for the 5MWT: for each walking-minute, 3 pain measurements will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* chronic nonspecific LBP for at least 3 months' duration: non-specific LBP implies that patients are not allowed to have any evidence of specific spinal pathology (e.g., hernia, spinal stenosis, spondylolisthesis, infection, spinal fracture or malignancy).

Exclusion Criteria:

* spinal surgery in the past 6 months
* severe underlying comorbidity (like diagnosed diabetes, cardiovascular problems, etc.),
* pregnant or given birth in the preceding year,
* having initiated a new LBP treatment in the 6 weeks prior to study participation

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Movement Evoked Pain | Change in pain score between (1) Movement Evoked Pain measures assessed without TENS application and (2) Movement-Evoked Pain measured assessed while using TENS application. Between both measures, a wash out period of 30 minutes was introduced.
  Pain that is experienced in response to 2 physical tasks: the Back Performance Scale and the 5 minutes walk test. Participants performed 5 physical tasks (= 1) grasping toes with fingertips in a sitting position; 2) forward bending from standing; 3) picking up paper from standing; 4) long-sitting from supine and 5) lifting a 5kg box from floor to table) and walked for 5 minutes. Participants provided a pain rating on a 11 points Numeric Rating Scale (NRS) with the endpoints no pain" (0) and "excruciating pain" (10). Pain will be assessed during the physical tasks (=at the same moment).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Leemans, Principal Investigator — Dra. Lynn Leemans
Locations (1):
- Vrije Universiteit Brussel, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

REFERENCES:
- [Background] Srikandarajah S, Gilron I. Systematic review of movement-evoked pain versus pain at rest in postsurgical clinical trials and meta-analyses: a fundamental distinction requiring standardized measurement. Pain. 2011 Aug;152(8):1734-1739. doi: 10.1016/j.pain.2011.02.008. Epub 2011 Mar 12. PMID 21402445